CLINICAL TRIAL: NCT05659030
Title: The Effect of Midwife-led Education Based on Pender's Health Promotion Model on Perinatal Mental Health of Migrant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Ayseren Cevik, Lecturer, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 04.11.2022/34
Record Dates: First submitted 2022-12-05; First posted 2022-12-21 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Mental Health; Perinatal Care
Keywords: Midwifery; human migration; mental health; perinatal care
MeSH Terms: conditions — Psychological Well-Being | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): It is planned to provide training on perinatal mental health to the experimental group in order to eliminate the lack of knowledge of women and to raise awareness. The pre-test will be applied during the pregnancy period before the training. These trainings, which will be held during pregnancy, consist of 3 modules. A training booklet in their preferred language (Turkish or Arabic) will be distributed to women at the end of each module. In addition, the effectiveness of the training will be evaluated at the end of each module and the knowledge deficiencies of women will be eliminated. A module training will be given every week and the training will be completed within three weeks. The effectiveness of the training will be evaluated in the postpartum period with the post-test.
  Interventions: Other: Education
- Control (No Intervention): Routine clinical care will be given to women in the control group. The pre-test will be applied during the pregnancy period and the post-test will be applied in the postpartum period. At the end of the post-test, three module training booklets will be distributed to the women in their preferred language (Turkish or Arabic). In line with their needs, the information deficiencies they request will be corrected.

INTERVENTIONS:
Other: Education — In order to develop the training material, first of all, a literature review will be made and a training booklet will be prepared. The training booklet will be submitted to expert opinion and a pilot application will be made by giving its final form. The training content is based on Pender's Health Promotion Model, which consists of 3 components.
  Arms: Experimental

SUMMARY:
This randomized controlled experimental study was conducted to evaluate the effects of midwife-led Pender's Health Promotion Model-based education given to immigrant women on perinatal mental health. The study was conducted with 52 intervention and 54 (n=48 in the post-test) control groups. The study consisted of five interviews. The intervention group received 3 modules of training, and the control group received routine clinical care.

DETAILED DESCRIPTION:
This randomized controlled experimental study was conducted to evaluate the effects of midwife-led Pender's Health Promotion Model-based education given to immigrant women on perinatal mental health. The study was conducted with 52 intervention and 54 (48 in the post-test) control groups. The study consisted of five interviews. Data were collected using an introductory information form, perinatal mental health information form, Edinburgh Postnatal Depression Scale and Perinatal Anxiety Screening Scale. Appropriate statistical analyses were performed in the analysis of data showing non-parametric distribution. The intervention group received 3 modules of training, and the control group received routine clinical care. The depression scores of the women in the intervention group did not show any significant difference over time, while the scores of the control group showed a significant difference. Depression scores between the groups showed significant differences in the third and fourth interviews. The anxiety scores of the women in the intervention and control groups showed a significant difference over time. No significant difference was observed between the groups in terms of anxiety scores. It can be said that the education based on Pender's Health Promotion Model has a protective and improving effect on perinatal health.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the study,
* Be over 18 years of age,
* Literate,
* Be of Syrian nationality and native Arabic,
* Be primiparous or multiparous,
* Be in the 28th-34th week of pregnancy.

Exclusion Criteria:

* Having a diagnosed risky pregnancy,
* Having a diagnosed mental illness (psychiatric report status, illness diagnosed by a psychiatrist and receiving treatment),
* Being benefited from psychological counseling, psychotherapy etc. services,
* Being excluded or excluded from the research at any stage of the research.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnancy
Enrollment: 106 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-12-09 (Actual)

PRIMARY OUTCOMES:
Perinatal Mental Health Education Evaluation Form | pre-intervention, immediately after the intervention, after 1 month.
  Change from the level of knowledge and awareness about perinatal mental health. An increase in the score is interpreted as an increase in the level of knowledge and awareness about perinatal mental.
Edinburgh Postnatal Depression Scale | pre-intervention, immediately after the intervention, after 1 month.
  Change from the prenatal and postnatal depression. An increase in the score is interpreted as an increase in perinatal depression symptoms. A score of 12 and above indicates the presence of depression.
Perinatal Anxiety Screening Scale | pre-intervention, immediately after the intervention, after 1 month.
  Change from prenatal and postnatal anxiety. An increase in the score is interpreted as an increase in perinatal anxiety symptoms. A score of 26 and above indicates the presence of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Ayseren Cevik, Msc, Principal Investigator — Cukurova University
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No